CLINICAL TRIAL: NCT06694220
Title: Impact of Tailored Preventive Exercise Program for Reducing Risk of Hip Adductors Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahinour Muhammed Osama, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PT REC/012/005100
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Adductor Strain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored preventive exercises and traditional exercises group (Experimental): The participants will practice tailored preventive exercises and traditional exercises for at least 6 weeks.
  Interventions: Other: Tailored preventive exercises; Other: Traditional exercises
- Traditional exercises group (Active Comparator): The participants will practice d traditional exercises for at least 6 weeks.
  Interventions: Other: Traditional exercises

INTERVENTIONS:
Other: Tailored preventive exercises — Players in the experimental group will be asked to perform the tailored preventive program 2-3 times per week for 1 hour for at least 6 weeks preseason which includes warming up for 10 mins, flexibility exercises, strengthening exercises, core and lower body stability and balance exercises and drills all these exercises for 1-4 sets x 10-20 reps and cooling down stretches for the last 10 mins.
  Arms: Tailored preventive exercises and traditional exercises group
Other: Traditional exercises — The players will be warmed up as usual, with jogging and ball-based exercises following FIFA 11+ warming up program which consist of three steps with 15 specific exercises running exercises for 8 mins, starting warming up in pairs; Path consists of 6-10 pairs of parallel cones: (Running Straight Ahead, Running Hip Out, Running Hip In, Running Circling Partner, Running Shoulder Contact, Running Quick Forwards and Backwards, Rep. x2). Strength, plyometric, balance for 10 minutes (The Bench, Sideways Bench, Single-leg Stance, Squats, Jumping Rep. 2x 30 sec each side). Running Exercises for 2 minutes (End of heating): (running across the pitch, running bounding, running plant, and cut. Rep x 2). Techniques need to be performed correctly and with an emphasis on maintaining the correct posture of the body. This exercise program should be done at least twice a week

SUMMARY:
this study will be conducted :

* To investigate the impact of tailored preventive exercise program in reducing hip adductor loss of isometric strength in professional football players.
* To investigate the impact of tailored preventive exercise program in reducing hip adductors to abductors strength asymmetry ratio in professional football players.
* To investigate the impact of tailored preventive exercise program in reducing pain intensity during seasonal matches in professional football players.
* To investigate the impact of tailored preventive exercise program on groin health and performance enhancement in professional football players.

DETAILED DESCRIPTION:
Football playing is associated with a high risk of injuries, which results in significant costs for the public health system and may even cause long-term disability for the injured player. The study's findings and the developed exercise program can have practical implications for athletic trainers, strength and conditioning coaches, and medical professionals working with professional football players. The program can serve as a valuable resource for designing individualized training regimens aimed at reducing adductor injury risk and optimizing performance in this specific sport population.

So, the study's significance lies in its focus on injury prevention programs, tailored training preventive programs, enhancing football players' performance on an evidence-based approach. Since there is still a lack of literature and a gap in this research area on the preventive exercise program related to sport injuries' field and as health care professionals, we must provide the best service for the players not only to increase their game performance but also to keep their long live journey of playing.

ELIGIBILITY:
Inclusion Criteria:

* Male football players only will be included in the study. Men's football had the second highest injury rates .
* Players will have loss in hip adductor strength more than 15% .
* Players will have hip adductor/abductor strength ratio in percent less than 80% or ratio less than 0.9.
* Participants will go under full documentation of groin health and injury history.
* Participants will Complain of muscle fatigue or spasm or mild pain on VAS will be 3 or less, during and after matches with no real injury.

Exclusion Criteria:

Presence of injuries at the level of the hip/hip region at the initial assessment

* Players with acute groin injuries.
* Players with recent hip and pelvic floor muscles problems.
* Players with acute hip adductor strains or tears.
* Players with inguinal hernia.
* Players who already don't play matches or stop training.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2025-02-10 (Estimated); Study Completion 2025-02-20 (Estimated)

PRIMARY OUTCOMES:
Isometric strength of hip adductor muscles | at least 6 weeks
  Isometric strength of hip adductor muscles of the dominant and non-dominant limb will be measured by hand held dynamometer (HHD) (Lafayette model 01165 manual muscle tester with 7 cm×3.5 cm pad) pre-season and post season.
  Players will be asked to complete a maximum repetition, pushing their distal shanks against the pads for 5 s, providing a measure of force (N) for left and right limbs. During testing, players will be allowed to hold the side of the plinths. The hip adductor strength test was performed three times, with a 45-second break between trials
Isometric asymmetry strength ratio between adductors and abductors | at least 6 weeks
  Isometric asymmetry strength ratio between adductors and abductors of dominant (kicking limb) and un-dominant limb (non-kicking limb) will be measured pre-season and post season using hand held dynamometer (HHD). Players will lay supine with the leg being tested in 0° hip and knee extension and resistance applied 5 cm proximal to the malleolus, while the leg not being tested was in knee flexion with the foot on the plinth.
Arabic version of Copenhagen HAGOS Questionnaire | at least 6 weeks
  HAGOS questionnaire will be evaluated pre-season and post season. It consists of 37 items covering 6 subscales (pain, symptoms, activities of daily living, sport and recreational activities, participation in physical activity, and quality of living and performance). Each scale from 0 to 4. The total is scored from 0 to 100 with a higher score indicating better hip and groin function.
Pain level | at least 6 weks
  Visual analogue scale will be used to measure pain level pre-season and post season. It is a 10 cm line with score ranged from 0 to 10. 0 indicates no pain and 10 indicates the worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Sohair shehata, Study Chair — Cairo University; Magda Ramadan, professor, Study Director — Cairo University
Locations (1):
- Mahinour muhammed osama, Cairo, Egypt